CLINICAL TRIAL: NCT03713424
Title: An fMRI Study of the Effects of Clavulanic Acid on Drug Addiction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Brett Froeliger, Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022247
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Clavulanic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clav (Active Comparator): 4-day 125 bid oral capsule administration
  Interventions: Drug: Clavulanic Acid
- Placebo (Placebo Comparator): 4-day, twice-daily oral capsule administration
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Clavulanic Acid — Beta lactamase inhibitor for smoking cessation
  Arms: Clav
Drug: Placebo oral capsule — placebo
  Arms: Placebo

SUMMARY:
This research study is looking into the effects of clavulanic on smoking behavior in adult cigarette smokers. The primary study hypothesis is that, compared to placebo, clavulanic acid will reduce smoking over the course of the study.

ELIGIBILITY:
Entry criteria:

Inclusion Criteria all subjects:

1. Age 18-65 years
2. English fluency
3. Functional vision (with corrective lenses as needed) to complete assigned assessments and tasks
4. Smoke > 10 cigarettes/day for a minimum of 2 yrs. and have an expired carbon monoxide (CO) concentration of ≥ 10 ppm (to confirm inhalation at screening and scanning)
5. If female, provide a negative urine pregnancy test.
6. Agrees to refrain from all other tobacco (i.e., dip/chew, cigars, cigarillos) and/or nicotine products (i.e., e-cigs, patches, gum/lozenges, inhalers/sprays) for the duration of study participation

Exclusion Criteria all subjects:

1. Sensitivity or allergy to clavulanic acid/antibiotics
2. Past head injury or primary neurological disorder associated with MRI abnormalities, including dementia, MCI, brain tumors, epilepsy, Parkinson's disease, or demyelinating diseases
3. Any physical or intellectual disability affecting completion of assessments
4. Any contraindication to MRI
5. Use of antidepressants medications with smoking cessation efficacy
6. Presence of an untreated illness or serious medical condition
7. Current or past psychosis
8. Electroconvulsive therapy in last 6 months
9. Positive pregnancy test (Urine pregnancy testing at screening and prior to fMRI scan) or currently breast feeding or BAC greater than 0.0
10. Use of carbamazepine or nitroglycerin (or any other medication deemed to be hazardous if taken with CLAV) within 14 days of study participation
11. Abnormal liver function determined by Complete Metabolic Panel - liver enzymes outside normal ranges of AST (SGOT) 5-40 unites/L and ALT( SGPT) 7-56units/L
12. Abnormal renal function determined by Complete Metabolic Panel - outside normal ranges of BUN 6-24 mg /dl and Creatinine level 0.6 -1.2 mg /dl male, 0.5-1.1mg /dl female
13. Any other condition or concern that in the investigator's opinion would impact participant safety, compliance with study instructions, or potentially confound the interpretation of the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-26 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Cigarette Smoking | 5 days
  Biochemical smoking assessment (breath carbon monoxide) at each study visit.
Self Reported Side Effects | 5 Days
  Number of reported side effects

SECONDARY OUTCOMES:
Magnitude of change in BOLD fMRI brain response to smoking related images | 4 days
  Measure the effects of Clavulanic Acid on fMRI BOLD response to images (change from baseline to end of study) while participants undergo functional magnetic resonance imaging
Magnitude of change in resting-stated fMRI brain connectivity | 4 days
  Measure the effects of Clavulanic Acid on resting-state functional connectivity (change from baseline to end of study) while participants undergo functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Froeliger, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri - Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No